CLINICAL TRIAL: NCT05614817
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Trial to Evaluate the Efficacy and Safety of CBP-201 Monotherapy in Patients With Moderate-To-Severe Atopic Dermatitis Who Are Candidates for Systemic Therapy
Brief Title: CBP-201 in Adolescent and Adult Patients With Moderate-to-severe Atopic Dermatitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-201-WW004; 2022-000999-19 (EudraCT Number)
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-01

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; allergic dermatitis; pruritis; type 2 inflammation; allergy
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- [Treatment Period 1]Group 1-Dose1 (Experimental): CBP-201 600 mg (4 mL) SC on Day 1 (Week 0 visit) visit followed by 300 mg (2 mL) SC Q2W starting at Week 2 with the last dose at Week 14.
  Interventions: Drug: CBP-201
- [Treatment Period 1]Goup 2-Placebo1 (Placebo Comparator): Placebo (4 mL) SC on Day 0 (Week 0) visit followed by placebo (2 mL) SC Q2W starting at Week 2 with the last dose at Week 14
  Interventions: Drug: Placebo
- [Treatment Period 2] Group 1-Dose2 (Experimental): CBP-201 300 mg SC Q2W starting at Week 16 with the last dose at Week 50 Treatment Period 2 (Group 1 Dose 1 responder pts that rerandomize to Dose 2, Dose 3, or PBO 2)
  Interventions: Drug: CBP-201
- [Treatment Period 2] Group 1-Dose3 (Experimental): CBP-201 300 mg SC Q4W starting at Week 16, alternating with placebo SC Q4W starting at Week 18 with the last dose of CBP-201 at Week 48 and placebo at Week 50
  Interventions: Drug: CBP-201
- [Treatment Period 2] Group 1-Placebo2 (Placebo Comparator): Placebo Q2W SC starting at Week 16 with the last dose at Week 50
  Interventions: Drug: Placebo
- [Treatment Period 2] Group 2-Placebo (Placebo Comparator): PBO 1 pts responders that continue PBO 1
  Interventions: Drug: Placebo
- [Treatment Period 2] Group 3-Dose (Experimental): Dose 1 and PBO 1 Non-responders, and Group 1 and 2 Non-responders that get open-label Dose 4 or 5 (LD 300 mg or 600 mg, biweekly 300 mg thereafter)
  Interventions: Drug: CBP-201

INTERVENTIONS:
Drug: CBP-201 — CBP-201 subcutaneous(SC) injection
  Arms: [Treatment Period 1]Group 1-Dose1; [Treatment Period 2] Group 1-Dose2; [Treatment Period 2] Group 1-Dose3; [Treatment Period 2] Group 3-Dose
Drug: Placebo — subcutaneous(SC) injection
  Arms: [Treatment Period 1]Goup 2-Placebo1; [Treatment Period 2] Group 1-Placebo2; [Treatment Period 2] Group 2-Placebo

SUMMARY:
This is a Phase 3, randomized, double-blinded, placebo-controlled trial in patients, ≥12 years of age who weigh ≥40 kg, and are diagnosed with moderate-to-severe AD.

DETAILED DESCRIPTION:
This study is comprised of a 2- to 6-week (Day-45 to Day 1) Screening Period, a 16-week randomized, double-blind Treatment Period 1, a 36-week Treatment Period 2, and an 8-week follow-up after the last dose of study drug. Therefore, participants will be enrolled in the trial for a maximum of 66 weeks.

ELIGIBILITY:
Inclusion Criteria:

-

* Able to provide written informed consent or assent (as per local law).
* Adults and adolescents of any sex or gender (12 years of age or older)
* Body weight ≥ 40 kg at Screening
* Diagnosis of chronic Atopic Dermatitis as defined according to American Academy of Dermatology Consensus Criteria (Eichenfield 2014), present ≥ 3 year before Screening.

Atopic Dermatitis history with ALL the following disease activity criteria:

1. Involvement of ≥ 10% BSA at Screening and Baseline (Day 1).
2. An EASI score of ≥ 16 at Screening and Baseline (Day 1).
3. An IGA score of ≥ 3 at Screening and Baseline (Day 1).
4. Baseline weekly average of daily PP-NRS ≥ 4 at Baseline (Day1).

   • Participant has applied a Sponsor approved emollient twice a day for at least 14 days before the Baseline Visit and agree to continue at least daily use during study participation.

   • Documented recent history (within 180 days before Screening) of inadequate response to treatment with TCS or topical immunomodulator medication or for whom topical treatments are otherwise medically inadvisable (e.g., important side effects or safety risks).
   * Participants must agree to avoid the use of prohibited AD medications throughout the duration of the study.
   * In the opinion of the Investigator, participant is willing and able to comply with all study visits and study-related procedures.
   * Female patients of childbearing potential who are sexually active with a non-sterilized male partner should have a confirmed negative serum beta-human chorionic gonadotropin test at Visit 1 and agrees to use acceptable forms of birth control.

Exclusion Criteria:

-

No current or past history of:

1. Other active skin diseases (e.g., psoriasis, lupus erythematosus etc.) or skin infections (bacterial, fungal, or viral) that require systemic treatment within 4 weeks of Screening Visit or would interfere with the assessment of AD lesions.
2. History of recurrent herpes herpeticum in the prior 12 months or more than 2 episodes of herpes herpeticum in past 2 years.
3. Non-skin related active infection requiring systemic treatment with parenteral anti-infectives within 30 days or oral anti-infectives within 14 days before the Baseline Visit (Visit 2).
4. Active human immunodeficiency virus (HIV) defined as a confirmed positive anti-HIV antibody test.
5. Tuberculosis requiring treatment within the past 12 months before Screening. Note: Evaluation of tuberculosis will be according to local guidelines as per standard of care.
6. Active Hepatitis B virus (HBV) or hepatitis C virus (HCV).
7. HCV: HCV ribonucleic acid (RNA) detectable in any subject with anti-HCV antibody (HCV Ab).

   •

Participant may not have any of the following conditions:

1. Known primary immunodeficiency or immunocompromised
2. History of malignancy within 5 years before the Screening Visit except for completely treated in situ carcinoma of the cervix or completely treated and resolved basal cell carcinoma of the skin.
3. A helminth parasitic infection diagnosed within 6 months before Visit 1 that has not been treated with or has failed to respond to standard of care therapy.
4. History of chronic alcohol or drug abuse including chronic use of cannabis (e.g., inhalation and/or consumption of marijuana more than once per week) within 12 months before screening.
5. History of attempted suicide or is at significant risk of suicide.
6. History of anaphylaxis after administration of a biologic medication or vaccine.
7. History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, e.g., monoclonal antibody) or to any of the study drug excipients [L-histidine, trehalose, or Tween (polysorbate) 80].
8. Any disorder, including, but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could: affect participant safety, alter the findings of the study or the interpretation of study results, impede the participant's ability to complete the entire duration of the study, or would require frequent bursts of systemic corticosteroids.

   * Participant may not have Prior/Concomitant Therapy as follows:

a. Receipt of live (attenuated) vaccines within 30 days of Baseline (Day 1) NOTE: Receipt of inactive/killed vaccines (e.g., influenza) or mRNA vaccines (e.g., COVID) are permitted provided that they are not given within 5 days before/after any of the study visits.

b. Receipt or donation of any blood product in the 28 days before Baseline (Day 1).

NOTE: Patients who are not willing to abstain from donating blood and/or plasma from Screening and for the 112 days after last dose of study drug should not be enrolled.

•

Participant is unable or unwilling to discontinue current prohibited AD treatments within defined washout windows below and in prohibited medications Section 6.11, as applicable, before Baseline (Visit 2):

1. Systemic JAK inhibitors including but not limited to ruxolitinib, tofacitinib, baricitinib, upadacitinib, abrocitinib and filgotinib within 60 days
2. Lymphocyte depleting agents such as rituximab within 6 months or when lymphocyte counts return to normal whichever is longer
3. Systemic therapy for AD including but not limited to corticosteroids, methotrexate, cyclosporine, azathioprine, phosphodiesterase type 4 (PDE-4) inhibitors, or mycophenolate mofetil within 4 weeks
4. Targeted biologic treatments (as listed in prohibited medication Section 6.11) within 5 half-lives (if known) or 12 weeks, whichever is longer
5. At any time prior to baseline, patient did not respond favorably to previous dupilumab or other anti-IL4Rα or anti-IL-13 treatment (e.g., therapy failure, patient experienced an adverse reaction to treatment)
6. Oral or parenteral traditional Chinese medicine within 4 weeks
7. Topical treatments other than the Sponsor permitted emollient, including but not limited to TCS, TCI, PDE-4, antihistamines, or JAKi within 2 weeks
8. Phototherapy treatment, laser therapy, tanning booth, or extended sun exposure that could affect disease severity or interfere with disease assessments within 4 weeks
9. Use of bleach baths in the prior 2 weeks
10. Topical anti-infectives within 2 weeks
11. Emollients only available by prescription within 2 weeks including those containing ceramide, hyaluronic acid, urea, filaggrin, Vitamin D or Vitamin E, even if not prescribed Prior/Concurrent Clinical Study Experience

    * Receipt of any experimental systemic medications in the 42 days before Baseline (Day 1), or 5 half-lives (if known), whichever is longer.
    * Previous enrollment in a CBP-201 treatment protocol and having received at least 1 dose of active study drug.
    * Concurrent enrollment in another trial where the patient is receiving an experimental intervention.

Have the following laboratory abnormalities at Screening:

1. Hemoglobin ≤ 10 g/dL
2. Platelet count < 100,000 cells/µL
3. Eosinophil count > 1500 cells/ µL
4. Total creatine phosphokinase (CPK) > 3 times the upper limit of the normal (ULN)
5. Alanine aminotransferase (ALT) ≥ 2.0xULN
6. Aspartate aminotransferase (AST) ≥ 2.0x ULN
7. Total Bilirubin ≥ 1.5x ULN (an isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated, and the direct bilirubin is < 35% or if the participant has known Gilbert's Syndrome)
8. Alkaline Phosphatase >2x ULN

   * Abnormal ECG at screening per investigator assessment.
   * Major surgery, requiring anesthesia, within 6 weeks before Baseline (Day 1), or planned in-patient surgery or hospitalization during study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Investigator Global Assessment(IGA)(0-1) | Baseline to Week16
  The proportion of participants whose IGA score is 0-1 and decreased by ≥2 points
EASI-75 | Baseline at Week 16
  The proportion of participants achieving EASI-75

SECONDARY OUTCOMES:
Change in Peak Pruritus Numerical Rating Scale（PP-NRS）(in the US) | Baseline at Week16
  The proportion of participants achieving an improvement (reduction) of ≥4 on Peak Pruritis numeric rating scale (PP-NRS)
Investigator Global Assessment(IGA)(0-1) (outside of the US) | Baseline at Week16
  Proportion of participants achieving an IGA score of 0 or 1 and a 2-grade improvement in IGA
Change in Peak Pruritus Numerical Rating Scale（PP-NRS）(outside of the US) | Baseline at Week16
  Proportion of participants achieving an improvement (reduction) of ≥4 on PP-NRS
Scoring Atopic Dermatitis(outside of the US) | At Week16
  Change in Scoring Atopic Dermatitis (SCORAD)
Dermatology Life Quality Index(outside of the US) | Baseline at Week16
  Change in Dermatology Life Quality Index (DLQI) score
EASI-90 | Baseline at Week16
  Proportion of participants achieving 90% reduction in EASI score

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC